CLINICAL TRIAL: NCT04993755
Title: A Phase 2a Study of TPN-101 in Patients With Amyotrophic Lateral Sclerosis (ALS) and/or Frontotemporal Dementia (FTD) Associated With Hexanucleotide Repeat Expansion in the C9orf72 Gene (C9ORF72 ALS/FTD)
Brief Title: A Phase 2a Study of TPN-101 in Patients With C9ORF72 ALS/FTD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Transposon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPN-101-C9-201
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontotemporal Dementia
Keywords: ALS; FTD
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TPN-101, 400 mg/day (Experimental)
  Interventions: Drug: TPN-101, 400 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TPN-101, 400 mg/day — 400 mg/day of study investigational drug TPN-101 once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: TPN-101, 400 mg/day
Drug: Placebo — Placebo once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to assess the the safety and tolerability of TPN-101 in patients with Amyotrophic Lateral Sclerosis (ALS) and/or Frontotemporal Dementia (FTD) Associated with Hexanucleotide Repeat Expansion in the C9orf72 gene (C9ORF72 ALS/FTD).

DETAILED DESCRIPTION:
This is a Phase 2a multi-center, randomized, double-blind, placebo-controlled parallel-group, 2-arm study with a long-term, open-label treatment phase in patients with C9ORF72 ALS and/or FTD. This study includes a 6-week Screening Period, a 24-week Double-blind Treatment Period, a 24-week Open-label Treatment Period, and a Follow-up Visit 4 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a clinical genetic test demonstrating a hexanucleotide repeat expansion (HRE) in the C9orf72 gene
* Has a reliable caregiver/informant to accompany the patient to all study visits

For patients with ALS (with or without FTD):

* Diagnosis of ALS (probable, possible, laboratory-supported probable or definite) according to the World Federation of Neurology revised E1 Escorial criteria
* Onset of weakness within 3 years prior to Screening
* Slow vital capacity (SVC) ≥ 60% of predicted normal adjusted for sex, age, and height (from the sitting position)
* Able to perform reproducible pulmonary function tests.
* ALS Functional Rating Scale-Revised (ALSFRS-R) ≥ 30 and score of 3 or 4 on Item #3 (swallowing) at Screening

For patients with FTD:

* A gradual, progressive decline in behavior, language, or motor function consistent with mild cognitive impairment, mild behavioral impairment, mild cognitive/behavioral impairment, behavioral variant FTD, primary progressive aphasia, or amnestic syndrome
* CDR Dementia Staging Instrument plus National Alzheimer's Coordinating Center Behavior and Language Domains (CDR plus NACC FTLD) global score of 0.5-2.0 at Screening

Exclusion Criteria:

* Presence of other significant neurological or psychiatric disorders
* History of clinically significant brain abnormality
* Clinically significant medical illness
* Tracheostomy or diaphragmatic pacing
* Autoimmune disease requiring treatment or management (quiescent rheumatoid arthritis, psoriasis, or controlled Type 1 diabetes are acceptable)
* History of human immunodeficiency virus (HIV) or hepatitis B infection, or any active infection during Screening, unless the patient will have been symptom-free for at least 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of TPN-101 in patients with C9ORF72 amyotrophic lateral sclerosis (ALS)/frontotemporal dementia (FTD) | 48 weeks
  Incidence and severity of spontaneously reported treatment-emergent adverse events (TEAEs) associated with TPN-101 v. placebo administered for up to 48 weeks in patients with C9ORF72 ALS/FTD

SECONDARY OUTCOMES:
Assess the pharmacokinetics of TPN-101 as measured by concentrations of TPN-101 in plasma and cerebrospinal fluid (CSF) | 48 weeks
Assess the pharmacodynamic effect of TPN-101 on neurodegeneration as measured by changes in the levels of CSF and blood neurofilament light (NfL) | 48 weeks
Assess the clinical effect of TPN-101 as measured by changes in score on the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 48 weeks
  The ALSFRS-R measures speech, salivation, swallowing, handwriting, cutting food and handling utensils (with or without gastrostomy), dressing and hygiene, turning in bed and adjusting bed clothes, walking, climbing, stairs, and breathing. Scores range from 0 to 40, with higher scores indicating that more function is retained.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (10):
  - University of California San Diego, La Jolla, California
  - University of California Irvine - ALS & Neuromuscular Center, Orange, California
  - UCSF Neurosciences Clinical Research Unit (NCRU), San Francisco, California
  - John Hopkins University, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Massachusetts General Hospital (MGH) - Amyotrophic Lateral Sclerosis (ALS) Multidisciplinary Clinic, Boston, Massachusetts
  - Mayo Family Clinic Northwest, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center - The Neurological Institute of New York, New York, New York
  - The University of North Carolina at Chapel Hill, Department of Neurology, Chapel Hill, North Carolina
- VIB-KU Leuven Center for Brain & Disease Research, Leuven, Flemish Brabankt, Belgium
- France (3):
  - CHU Lille - CMRR Hôpital Roger Salengro, Lille
  - CHU Dupuytren, Limoges, Limoges
  - Groupe Hospitalier Pitie-Salpetriere - La Federation de Maladies du Systeme Nerveux, Paris
- Universitaetsklinikum Ulm - Klinik fuer Neurologie, Ulm, Baden-Wurttemberg, Germany
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari I Politècnic La Fe, Valencia